CLINICAL TRIAL: NCT06609226
Title: An Open-label, Multi-centre, Rollover Study to Characterise Long-term Safety and Efficacy of Etavopivat in Adults, Adolescents and Children Who Have Sickle Cell Disease or Thalassaemia and Have Completed a Treatment Period in an Etavopivat Study
Brief Title: A Research Study Looking at Long-term Treatment With Etavopivat in People With Sickle Cell Disease or Thalassaemia
Acronym: FLORAL
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN7535-7822; U1111-1301-8130 (Other: Universal Trial Number); 2024-510805-27 (Other: EU CT Number)
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Sickle Cell Disease; Thalassemia
MeSH Terms: conditions — Anemia, Sickle Cell; Thalassemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Participants greater than or equal to (≥) 12 years old with sickle cell disease (Experimental): Participants will receive an oral dose of Etavopivat A or C.
  Interventions: Drug: Etavopivat A; Drug: Etavopivat C
- Participants ≥ 12 years old with sickle cell disease transfusion dependent (Experimental): Participants will receive an oral dose of Etavopivat A or C.
  Interventions: Drug: Etavopivat A; Drug: Etavopivat C
- Participants ≥ 12 years old with transfusion-dependent thalassaemia (Experimental): Participants will receive an oral dose of Etavopivat A or C.
  Interventions: Drug: Etavopivat A; Drug: Etavopivat C
- Participants ≥ 12 years old with non-transfusion dependent thalassaemia (Experimental): Participants will receive an oral dose of Etavopivat A or C.
  Interventions: Drug: Etavopivat A; Drug: Etavopivat C
- Participants ≥ 2 years to less than (<) 12 years old with sickle cell disease (Experimental): Participants ≥ 12 years of age will receive an oral dose of Etavopivat A or C and participants < 12 years of age will receive an oral dose of Etavopivat B.
  Interventions: Drug: Etavopivat A; Drug: Etavopivat B; Drug: Etavopivat C

INTERVENTIONS:
Drug: Etavopivat A — Participants will receive an oral dose of Etavopivat A.
Drug: Etavopivat B — Participants will receive an oral dose of Etavopivat B.
  Arms: Participants ≥ 2 years to less than (<) 12 years old with sickle cell disease
Drug: Etavopivat C — Participants will receive an oral dose of Etavopivat C.

SUMMARY:
Etavopivat is a new medicine under development for treating blood disorders like sickle cell disease and thalassaemia. Sickle cell disease and thalassaemia are inherited blood disorders that affect haemoglobin. Haemoglobin is the protein that carries oxygen through the body. This study is looking into how safe treatment with etavopivat is and how well it works over a long period of time. The study will last for up to 264 weeks, but it will end earlier if etavopivat is approved in the participant's country.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have ongoing participation in an etavopivat parent study for treatment of sickle cell disease (SCD) or thalassaemia and have completed at least a treatment period of the parent study.
* Participant must have derived clinical benefit from treatment with etavopivat, as determined by the investigator.
* Any participant with dose reduction or temporary discontinuation will need to be successfully rechallenged to the full dose of etavopivat before transferring.
* Participants on hydroxyurea (HU), crizanlizumab or l-glutamine oral powder (Endari®) treatment at the time of consent may be eligible if they have been on a stable dose in the parent study as defined at the investigator's discretion. Necessary adjustments related to weight or age are accepted. Participants with temporary dose reductions or pauses due to medical reasons may still be considered to have a stable dose, as determined by the investigator, who will assess the impact of these adjustments based on clinical context and the participant's overall health status.

Exclusion Criteria:

* Any disorder, except for conditions associated with SCD or thalassaemia, which in the investigator's opinion might jeopardise participant's safety or compliance with the protocol.
* Participant withdrew or had permanent treatment discontinuation from an etavopivat clinical study.
* Participants on permanent dose reduction (greater than [>] 28 days or more) or ongoing temporary treatment discontinuation.
* Use of any of the following within the timeframes prior to the transfer visit as stated:
* Use of haemoglobin S (HbS) polymerisation inhibitors within participation of the parent study or anticipated need for this agent during this study.
* Use of an experimental selectin antagonist (e.g., monoclonal antibody or small molecule) within the parent study or anticipated need for such agents during this study.
* Use of erythropoietin or other haematopoietic growth factor treatment for more than 4 consecutive weeks during the parent study or anticipated need of such agents for a maintenance treatment during this study.
* Receiving or use of concomitant medications that are strong inducers of cytochrome P450 (CYP) 3A4 within 2 weeks of the transfer visit or anticipated need for such agents during the study.
* Current participation in a study that is not a designated parent study, or planned participation in any other clinical study, for the duration of FLORAL.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2030-12-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events (TEAEs), reported for each indication and age group separately | Baseline (week 0 of FLORAL) up to end of study (up to week 316)
  Measured as number of events.
Number of adverse reactions, reported for each indication and age group separately | Baseline (week 0 of FLORAL) up to end of study (up to week 316)
  Measured as number of adverse reactions.

SECONDARY OUTCOMES:
Annualised vaso-occlusive crisis (VOC) rates, reported for each age group separately | Baseline (week 0 of FLORAL) up to end of treatment (up to week 312)
  Measured as count.
Change in VOCs, reported for each age group separately | Baseline (of parent study [i.e., the previous etavopivat study that a participant is rolling over from]) up to end of treatment (up to week 312)
  Measured as count.
Change in hemoglobin (Hb) concentration, reported for each age group separately | Baseline (of parent study [i.e., the previous etavopivat study that a participant is rolling over from]) up to end of treatment (up to week 312)
  Measured as grams per deciliter (g/dL).
Annualised number of hospitalisations, reported for each age group separately | Baseline (week 0 of FLORAL) up to end of treatment (up to week 312)
  Measured as count.
Average length of stay of hospitalisations, reported for each age group separately | Baseline (week 0 of FLORAL) up to end of treatment (up to week 312)
  Measured as days.
Change in Hb concentration | Baseline (of parent study [i.e., the previous etavopivat study that a participant is rolling over from]) up to end of treatment (up to week 312)
  Measured as g/dL.
Number of red blood cell (RBC) units transfused, reported for each indication separately | Baseline (week 0 of FLORAL) up to end of treatment (up to week 312)
  Measured as units.
Change in RBC units transfused, reported for each indication separately | Baseline (of parent study [i.e., the previous etavopivat study that a participant is rolling over from]) up to end of treatment (up to week 312)
  Measured as units.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (99):
- United States (36):
  - Univ of Alabama Birmingham, Birmingham, Alabama
  - Phoenix Children's Hsptl, Phoenix, Arizona
  - Children's Hospital Los Angeles - Endocrinology, Los Angeles, California
  - UCSF Oakland Benioff ChildHosp, Oakland, California
  - Children's Hosp Of Orange, Orange, California
  - University Of California Irvine, Orange, California
  - University of Connecticut, Farmington, Connecticut
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Foundation for Sickle Cell Disease Research, Hollywood, Florida
  - Univ of Miami/SCCC, Miami, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Children's Healthcare Atlanta, Atlanta, Georgia
  - Center for Blood Disorders Augusta University, Augusta, Georgia
  - Univer Of Illinois at Chicago, Chicago, Illinois
  - Children's Hosp-New Orleans, New Orleans, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Washington University-St.Louis, St Louis, Missouri
  - NYC Health+Hospitals, Brooklyn, New York
  - Columbia University Medical Center_New York_0, New York, New York
  - Weill Cornell Med Coll-NYPH, New York, New York
  - Jacobi Medical Center, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York
  - Atrium Levine Children's/Atrium Health, Charlotte, North Carolina
  - Duke University_Durham, Durham, North Carolina
  - East Carolina Univ-Greenville, Greenville, North Carolina
  - East Carolina University_Greenville, Greenville, North Carolina
  - Atrium Health-Wake Forest Bapt, Winston-Salem, North Carolina
  - Cincinnati Child's Hsp Med Ctr, Cincinnati, Ohio
  - Neuro-Behavioral Clinical Research, North Canton, Ohio
  - Medical University Of South Carolina_Charleston, Charleston, South Carolina
  - Methodist University Hospital, Memphis, Tennessee
  - Texas Children's Hospital_Houston, Houston, Texas
  - UT Health University of Texas, Houston, Texas
  - Virginia Comm Univ Medical Ctr, Richmond, Virginia
  - Mary Bridge Children's Health, Tacoma, Washington
  - Versiti, CCBD_Milwaukee, Milwaukee, Wisconsin
- Canada (4):
  - St Pauls Hospital, Vancouver, British Columbia
  - The Hospital for Sick Children, Toronto, Ontario
  - University Health Network - Toronto General Hospital, Toronto, Ontario
  - CHU Ste-Justine, Montreal, Quebec
- Egypt (5):
  - Alexandria University Hospital, Alexandria, Egypt
  - Zagazig University Hospital, Alsharkia, Egypt
  - Faculty of Medicine Ain Shams Medical Research Institute (MASRI), Cairo
  - Cairo University, Cairo, Egypt
  - Abu El-Reesh El-Mounira Children University Hospital, Cairo, Egypt
- France (3):
  - Ap-Hp-Hopital Henri Mondor, Créteil
  - Hospices Civils de Lyon-Hopital Edouard Herriot, Lyon
  - Ap-Hp-Hopital Robert Debre, Paris
- Germany (2):
  - Charité - Campus Virchow-Klinikum - Klinik für Pädiatrie mit Schwerpunkt Onkologie und Hämatologie, Berlin
  - Universitätsklinikum Freiburg - Kinder- und Jugendklinik, Freiburg im Breisgau
- Ghana (2):
  - Kintampo Health Research Centre (KHRC), Kintampo, Bono East
  - Ghana Institute of Clinical Genetics, Korle Bu Teaching Hospital (KBTH), Accra
- Greece (4):
  - General Hospital Of Larissa Koutlibaneio And Triantafylleio - Thalassemia and SCD Unit, Larissa, Thessaly
  - Hippokration Hospital, Athens
  - General University Hospital of Patras, Pátrai
  - 'Ippokrateio' General Hospital of Thessaloniki, Thessaloniki
- India (6):
  - All India Institute of Medical Sciences (AIIMS), Raipur, Raipur, Chhattisgarh
  - K.J Somaiya Hospital and Research Centre, Mumbai, Maharashtra
  - Victoria Hospital, Bangalore, Bangalore
  - Nirmal Hospital Pvt. Ltd., Gujarat
  - Suretech Hospital and Research Centre Ltd., Maharashtra
  - All India Institute of Medical Sciences_Delhi, New Delhi
- Italy (3):
  - Azienda Ospedaliera Universitaria San Luigi Gonzaga - S.C.D.O. Microcitemie e malattie rare ematologiche, Orbassano, Torino
  - Azienda Ospedale Universita Padova, Padua
  - Fondazione IRCCS Policlinico San Matteo, Pavia
- Kenya (6):
  - Gertrude's Children's Hospital, Nairobi, Nairobi County
  - KEMRI CRDR Siaya Clinical Research Annex, Country Referral Hospital, Siaya, Siaya County
  - KEMRI-Walter-Reed Kericho, Kericho
  - Kombewa Clinical Research Centre, Kisumu
  - KEMRI Kondele Children Hospital, Kisumu, Kisumu
  - Ahero Clinical Trials Unit, Kisumu
- Lebanon (3):
  - American University of Beirut Medical Centre, Hamra
  - Chronic Care Center, Hazmiyeh
  - Hospital Nini, Tripoli
- Nigeria (6):
  - University of Nigeria Teaching Hospital (UNTH), Ituku-Ozalla, Enugu State
  - University College Hospital Paediatric Haematology and Oncology Unit, Ibadan, Ibadan, Oyo State
  - University of Abuja Teaching Hospital, Gwagwalada, Abuja, Abuja
  - Barau Dikko Teaching Hospital, Kaduna, Kaduna
  - Aminu Kano Teaching Hospital (AKTH), Kano
  - Lagos University Teaching Hospital, Lagos, Lagos
- Sultan Qaboos University Hospital, Muscat, Sultanet of Oman/Muscat/Al Khoud, Oman
- Saudi Arabia (2):
  - Prince Mohammad Bin Naser Hospital, Jizan
  - King Khalid University Hospital, Riyadh
- Spain (3):
  - Hospital Universitario de Cruces, Barakaldo
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Universitario La Paz, Madrid
- Turkey (Türkiye) (6):
  - Baskent Universitesi Adana, Adana
  - Başkent Üniversitesi Adana-Hematoloji, Adana
  - Hacettepe University Hematology, Ankara
  - Hacettepe Üniversitesi Hastanesi- Hematoloji, Ankara
  - Mersin University Medical Faculty Pediatric Hematology, Mersin
  - Mersin Üniversitesi Tip Fakültesi Hastanesi- Çiftlikköy Yerleşkesi- Hematoloji, Mersin
- United Kingdom (7):
  - Guy's Hospital - Haematology, London
  - Guy's Hospital, London
  - King's College Hospital - Paediatric Research, London
  - Kings College Hospital - Haematology, London
  - Imperial College London, London
  - Manchester Royal Infirmary, Manchester
  - Royal Hallamshire Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com